CLINICAL TRIAL: NCT02565173
Title: Phase III Multi-center, Randomized, Double-masked, Active- and Placebo-controlled Study of Trabodenoson in Adults With Ocular Hypertension or Primary Open-angle Glaucoma
Brief Title: Study of Trabodenoson in Adults With Ocular Hypertension or Primary Open-angle Glaucoma
Acronym: MATrX-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Inotek Pharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IPC-01-2015
Record Dates: First submitted 2015-09-28; First posted 2015-10-01 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Primary Open-Angle Glaucoma (POAG); Ocular Hypertension (OHT)
Keywords: glaucoma; primary open-angle glaucoma; ocular hypertension; adenosine agonist; eye drop; trabodenoson; trabecular meshwork
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — trabodenoson; BID protein, human; INO-8875; Timolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- trabodenoson 4.5% BID (Experimental): trabodenoson 4.5% Ophthalmic Formulation
  Interventions: Drug: trabodenoson 4.5% BID
- trabodenoson 6.0% QD (Experimental): trabodenoson 6.0% Ophthalmic Formulation
  Interventions: Drug: trabodenoson 6.0% QD
- trabodenoson 3.0% QD (Experimental): trabodenoson 3.0% Ophthalmic Formulation
  Interventions: Drug: trabodenoson 3.0% QD
- timolol 0.5% BID (Active Comparator): timolol 0.5% Ophthalmic Formulation
  Interventions: Drug: timolol 0.5% BID
- placebo BID (Placebo Comparator): placebo Ophthalmic Formulation
  Interventions: Drug: placebo BID

INTERVENTIONS:
Drug: trabodenoson 4.5% BID — Trabodenoson 4.5% administered twice per day in both eyes for 12 weeks.
  Other Names: INO-8875
  Arms: trabodenoson 4.5% BID
Drug: trabodenoson 6.0% QD — Trabodenoson 6.0% administered once per day in the morning in both eyes followed by matching placebo administered once per day in the evening in both eyes for 12 weeks.
  Other Names: INO-8875
  Arms: trabodenoson 6.0% QD
Drug: trabodenoson 3.0% QD — Trabodenoson 3.0% administered once per day in the morning in both eyes followed by matching placebo administered once per day in the evening in both eyes for 12 weeks.
  Other Names: INO-8875
  Arms: trabodenoson 3.0% QD
Drug: timolol 0.5% BID — Timolol 0.5% administered twice per day in both eyes for 12 weeks.
  Other Names: Timoptic
  Arms: timolol 0.5% BID
Drug: placebo BID — Placebo administered twice per day in both eyes for 12 weeks.
  Arms: placebo BID

SUMMARY:
Phase III trial involving topical application, in both eyes, of trabodenoson ophthalmic formulation 3.0% or 6.0% once per day or 4.5% twice per day, placebo twice per day, or timolol 0.5% twice per day for 12 weeks in adult subjects with Ocular Hypertension or Primary Open-Angle Glaucoma.

All subjects who meet the study's enrollment criteria following Screening will undergo washout of all prohibited medications, including their routine glaucoma medications. During the Placebo Run-In Period, placebo is administered twice daily to both eyes in all subjects. During the Treatment Period, study drug is applied to both eyes for a total of 12 weeks followed by an Observation Period of approximately 7 days wherein no study eye drops are instilled.

The purpose of the study is to assess the efficacy, tolerability, and safety of binocular topical application of trabodenoson ophthalmic formulation 3.0% or 6.0% QD or 4.5% BID for 12 weeks.

Timolol is being included in the trial in order to have an active control to ensure the integrity of the trial from an efficacy perspective; the primary comparator for all statistical purposes is the placebo arm.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ocular hypertension (OHT) or primary open-angle glaucoma (POAG)
* Mean Intraocular pressure (IOP) of ≥24 and ≤34

Exclusion Criteria:

* Significant visual field loss or any new field loss within the past year
* Cup-to-disc ratio >0.8
* Central corneal thickness <490 µm or >610 µm
* A recent (acute) or chronic medical condition that might obfuscate the Subject's study data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2015-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Mean Intraocular Pressure (IOP) | Three Months

OTHER OUTCOMES:
Safety Parameters, including treatment emergent adverse events, to assess tolerability and safety. | Through Study Completion, up to 13 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Cadmus C Rich, MD,MBA,CPE, Study Director — Inotek Pharmaceuticals Corp.
Locations (1):
- Inotek Pharmaceuticals Corporation, Lexington, Massachusetts, United States